CLINICAL TRIAL: NCT00472290
Title: An Open Label Extension Study Evaluating the Safety of Long Term Dosing of Romiplostim in Thrombocytopenic Subjects With Myelodysplastic Syndromes (MDS)
Brief Title: Evaluating the Safety of Long Term Dosing of Romiplostim (Formerly AMG 531) in Thrombocytopenic Subjects With Myelodysplastic Syndromes (MDS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20060197
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Results first posted 2013-07-15 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Hematology; MDS; Myelodysplastic Syndromes; Thrombocytopenia
Keywords: Hematology; MDS; Myelodysplastic Syndromes; Thrombocytopenia
MeSH Terms: conditions — Myelodysplastic Syndromes; Thrombocytopenia | interventions — romiplostim

ARMS (1):
- Open Label Romiplostim (formerly AMG 531) (Experimental)
  Interventions: Drug: Romiplostim (formerly AMG 531)

INTERVENTIONS:
Drug: Romiplostim (formerly AMG 531) — Subjects will begin the study at an initial dose of 750 µg.
  Except for:
  * Subject whose doses were escalated to doses higher than 750 µg AMG 531 weekly, and maintained a response per IWG guidelines for platelet response.
  * Subjects who were stable at a lower dose of AMG 531 on the previous study. Doses will be adjusted throughout the study based on individual subject's platelet count.

SUMMARY:
This is an open label extension study of romiplostim for treatment of thrombocytopenia (platelet count ≤ 50 x 10^9/L) in MDS subjects. The study is designed to assess the long-term safety of treatment with romiplostim, as measured by incidence of overall adverse events, the incidence of bleeding events, the utilization of platelet transfusions, and the duration of platelet response. The study will further describe the time to disease progression to acute myeloid leukemia (AML) and survival.

ELIGIBILITY:
Inclusion Criteria

* Subject completed a romiplostim study for the treatment of thrombocytopenia in subjects with MDS
* Subject has an Eastern Cooperative Oncology (ECOG) performance status of 0 to 2
* Subject had a platelet count ≤ 50 x 10^9/L since the final dose of investigational product in the parent study
* Subject or his/her legally acceptable representative provided written informed consent before any study-specific procedures were initiated

Exclusion Criteria

* Subject has been diagnosed with AML or has a blast count ≥ 10% by peripheral blood or bone marrow biopsy
* Subject has a prior history of leukemia
* Subject has a prior history of bone marrow or stem cell transplantation
* Subject has a prior malignancy (other than in situ cervical cancer, controlled prostate cancer, or basal cell cancer of the skin) unless treated with curative intent and without evidence of disease for ≥ 3 years before randomization
* Subject has active or uncontrolled infections
* Subject has unstable angina, congestive heart failure [New York Heart Association (NYHA) > class II], uncontrolled hypertension (diastolic > 100 mmHg), uncontrolled cardiac arrhythmia, or recent (within 1 year) myocardial infarction
* Subject has a history of arterial thrombosis (eg, stroke or transient ischemic attack) in the past year
* Subject has a history of venous thrombosis that currently requires anti-coagulation therapy
* Subject received interleukin (IL)-11 within 4 weeks of screening
* Subject previously received a thrombopoietic growth factor (other than romiplostim)
* Subject has a known hypersensitivity to any recombinant E coli-derived product (eg, Infergen®, Neupogen®, Somatropin, Actimmune)
* Subject is currently enrolled in investigational device or drug study(ies), has not yet completed at least 4 weeks since ending investigational device or drug study(ies) (other than parent romiplostim study), or subject is receiving other investigational agent(s)/device(s)
* Subject is of child-bearing potential and is evidently pregnant (eg, positive human chorionic gonadotropin [HCG] test) or is breast feeding
* Subject is not using adequate contraceptive precautions
* Subject has any kind of disorder that compromises his/her ability to give written informed consent (and does not have a legally acceptable representative) or is unable to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2007-04-01 (Actual); Primary Completion 2011-07-18 (Actual); Study Completion 2011-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Derived] Fenaux P, Muus P, Kantarjian H, Lyons RM, Larson RA, Sekeres MA, Becker PS, Orejudos A, Franklin J. Romiplostim monotherapy in thrombocytopenic patients with myelodysplastic syndromes: long-term safety and efficacy. Br J Haematol. 2017 Sep;178(6):906-913. doi: 10.1111/bjh.14792. Epub 2017 Jun 14. PMID 28616874
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was available to subjects who completed a previous romiplostim study for the treatment of thrombocytopenia in subjects with low or intermediate-1 risk MDS. First Subject Enrolled: 17-Jul-2007; Last Subject Enrolled: 15-Feb-2011
Groups:
- Romiplostim: Subjects received subcutaneous dosing at 250, 500, 750, 1000, or 1500 mcg weekly or biweekly, with adjustments based on platelets. Romiplostim is supplied in a 5 mL single use vial as a sterile, white, preservative-free, lyophilized powder.
Period: Overall Study
Arm/Group | Romiplostim
Started | 72
Completed | 0
Not Completed | 72
Not completed — Progression of Therapy-Related MDS | 1
Not completed — Protocol Specified Criteria | 7
Not completed — Administrative Decision | 37
Not completed — Death | 3
Not completed — Lost to Follow-up | 1
Not completed — Lack of Efficacy | 1
Not completed — Disease Progression | 4
Not completed — Withdrawal by Subject | 5
Not completed — Adverse Event | 6
Not completed — Requirement for alternative therapy | 7

BASELINE CHARACTERISTICS:
Arm/Group | Romiplostim
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 40
Race/Ethnicity, Customized [Number; unit: Participant]
  White or Caucasian | 61
  Black or African American | 4
  Hispanic or Latino | 3
  Other | 4
Myelodysplastic Syndromes World Health Organization Classification at Study Screening [Number; unit: Participants]
  RA: Refractory Anemia | 20
  RARS: Refractory Anemia with Ringed Sideroblasts | 1
  RAEB-1: Refractory Anemia with Excess Blasts-1 | 7
  RAEB-2: Refractory Anemia with Excess Blasts-2 | 2
  RCMD:Refractory cytopenia w multilineage dysplasia | 24
  RCMD-RS: RCMD and ringed sideroblasts | 3
  MDS-U: Myelodysplastic syndrome - unclassified | 15
  MDS associated with isolated del(5q) | 0
Eastern Cooperative Oncology (ECOG) performance status [Number; unit: Participants]
  0: Fully active | 42
  1: Can carry out light or sedentary work | 25
  2: Capable of selfcare but unable to work | 5
  >=3: Capable of only limited selfcare or worse | 0
Baseline Platelet Count [Mean (Standard Deviation); unit: 10^9/L] | 27.6 (15.5)

OUTCOME MEASURES:

1. Primary Outcome: Overall Summary of Adverse Events
Time Frame: During treatment period from first dose of IP to End of Study visit, on Average 56 Weeks .
Population: Safety analysis includes subjects who took at least one dose of romiplostim.
Measure: Number; unit: Participant
Arm/Group | Romiplostim
Number analyzed (Participants) | 72
Participant
  Subjects Reporting Any AE | 71
  Subjects Reporting Any Treatment-related AE | 19
  Subjects Reporting Any Treat-related Serious AE | 4
  Subjects Reporting Any Serious AE | 29
  Subjects Withdrew Study or Stop IP Due to AE | 8

2. Secondary Outcome: Weekly Bleeding Events Per 100 Subject Years
Description: During the time since the first dose of IP to the end of the treatment period. A single bleeding event was defined as each individual bleeding episode that originated from a specific organ system (eg, gastrointestinal system or central nervous system). A bleeding event that continued for more than 7 days was counted as separate events every eighth day.
Time Frame: During the treatment period. The average duration of romiplostim exposure is 56 weeks.
Population: Safety analysis includes subjects who received at least one dose of romiplostim.
Measure: Mean (95% Confidence Interval); unit: Events/100 subject-year
Units Other Than Participants: Events
Arm/Group | Romiplostim
Number analyzed (Participants) | 72
Number analyzed (Events) | 866
Events/100 subject-year | 1120.5 [1047.1 to 1197.7]

3. Secondary Outcome: Platelet Transfusion Events Per 100 Subject Years
Description: During the time since the first dose of IP to the end of the treatment period. A discrete platelet transfusion event was defined as any number of platelet transfusions administered within a 3-day period. Platelet transfusions administered more than 3 days apart were counted as separate platelet transfusion events.
Time Frame: During the treatment period. The average duration of romiplostim exposure is 56 weeks.
Population: Safety analysis includes subjects who received at least one dose of romiplostim.
Measure: Mean (95% Confidence Interval); unit: Events/100 subject-year
Units Other Than Participants: Events
Arm/Group | Romiplostim
Number analyzed (Participants) | 72
Number analyzed (Events) | 158
Events/100 subject-year | 204.4 [173.8 to 238.9]

4. Secondary Outcome: Weeks With Platelet Response Per Year
Description: During the time since the first dose of IP to the end of the treatment period. Platelet response was based on the modified IWG 2006 criteria (Cheson et al, 2006) and was defined as, in the absence of platelet transfusion: an absolute increase in platelet count of ≥ 30 x 10^9/L for a subject starting with a platelet count of ≥ 20 x 10^9/L; or an increase in platelet count from < 20 x 10^9/L to ≥ 20 x 10^9/L and by at least 100% in a subject that started with a platelet count < 20 x 10^9/L.
Time Frame: During the treatment period. The average duration of romiplostim exposure is 56 weeks.
Population: Safety analysis includes subjects who received at least one dose of romiplostim.
Measure: Mean (95% Confidence Interval); unit: Weeks/Subject-year
Units Other Than Participants: Weeks with Platelet Response
Arm/Group | Romiplostim
Number analyzed (Participants) | 72
Number analyzed (Weeks with Platelet Response) | 2675
Weeks/Subject-year | 34.6 [33.3 to 35.9]

5. Secondary Outcome: Time to First Platelet Response
Description: Time since first dose of IP to the first platelet response. Platelet response was based on the modified IWG 2006 criteria (Cheson et al, 2006) and was defined as, in the absence of platelet transfusion: an absolute increase in platelet count of ≥ 30 x 10^9/L for a subject starting with a platelet count of ≥ 20 x 10^9/L; or an increase in platelet count from < 20 x 10^9/L to ≥ 20 x 10^9/L and by at least 100% in a subject that started with a platelet count < 20 x 10^9/L.
Time Frame: During treatment period. The average duration of romiplostim exposure is 56 weeks.
Population: Safety analysis includes subjects who received at least one dose of romiplostim.
Measure: Median (95% Confidence Interval); unit: Weeks
Units Other Than Participants: Weeks with Platelet Response
Arm/Group | Romiplostim
Number analyzed (Participants) | 72
Number analyzed (Weeks with Platelet Response) | 2675
Weeks | 2.3 [2.1 to 3.1]

6. Secondary Outcome: Duration of Platelet Response
Description: Platelet response was based on the modified IWG 2006 criteria (Cheson et al, 2006) and was defined as, in the absence of platelet transfusion: an absolute increase in platelet count of ≥ 30 x 10^9/L for a subject starting with a platelet count of ≥ 20 x 10^9/L; or an increase in platelet count from < 20 x 10^9/L to ≥ 20 x 10^9/L and by at least 100% in a subject that started with a platelet count < 20 x 10^9/L.
Time Frame: During treatment period. The average duration of romiplostim exposure is 56 weeks.
Population: Safety analysis includes subjects who received at least one dose of romiplostim.
Measure: Median (Full Range); unit: Weeks
Units Other Than Participants: Weeks with Platelet Response
Arm/Group | Romiplostim
Number analyzed (Participants) | 72
Number analyzed (Weeks with Platelet Response) | 2675
Weeks | 20.0 (49.5) [1 to 159]

7. Primary Outcome: Incidence of Antibody (AB) Formation
Time Frame: During treatment period from first dose of IP to End of Study visit, on Average 56 Weeks.
Population: Safety analysis includes subjects who took at least one dose of romiplostim.
Measure: Number; unit: Participant
Arm/Group | Romiplostim
Number analyzed (Participants) | 72
Participant
  Positive binding AB to IP at or before baseline | 5 (94.7)
  Neutralizing AB to IP at or before baseline | 0
  Binding AB positive to IP post-baseline only | 5
  Persistent binding AB positive to IP | 4
  Transient binding AB positive to IP | 1
  Positive binding AB to TPO at or before baseline | 4
  Neutralizing AB to TPO at or before baseline | 0
  Binding AB positive to TPO post-baseline only | 3
  Persistent binding AB positive to TPO | 2
  Transient binding AB positive to TPO | 1

ADVERSE EVENTS:
Time Frame: The average duration is 56 weeks
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Romiplostim
Serious Adverse Events (participants affected / at risk) | 29/72
Other Adverse Events (participants affected / at risk) | 66/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Romiplostim (N=72)
Anaemia (Blood and lymphatic system disorders) | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Muscular dystrophy (Congenital, familial and genetic disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Varices oesophageal (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chest pain (General disorders) | 1
Fatigue (General disorders) | 1
Pyrexia (General disorders) | 1
Bacteraemia (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 2
Diverticulitis (Infections and infestations) | 1
Fungaemia (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Fall (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Blood creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebral ischaemia (Nervous system disorders) | 1
Depressed level of consciousness (Nervous system disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Hepatic encephalopathy (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Speech disorder (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Renal failure acute (Renal and urinary disorders) | 2
Endometrial hypertrophy (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hilum mass (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary vascular disorder (Respiratory, thoracic and mediastinal disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Haematoma (Vascular disorders) | 3
Phlebitis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Romiplostim (N=72)
Anaemia (Blood and lymphatic system disorders) | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Palpitations (Cardiac disorders) | 4
Eye haemorrhage (Eye disorders) | 7
Abdominal pain (Gastrointestinal disorders) | 12
Constipation (Gastrointestinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 8
Gingival bleeding (Gastrointestinal disorders) | 8
Haemorrhoids (Gastrointestinal disorders) | 6
Mouth haemorrhage (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 6
Toothache (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 8
Asthenia (General disorders) | 6
Fatigue (General disorders) | 15
Oedema peripheral (General disorders) | 5
Pain (General disorders) | 6
Pyrexia (General disorders) | 9
Bronchitis (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 7
Sinusitis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 9
Urinary tract infection (Infections and infestations) | 6
Contusion (Injury, poisoning and procedural complications) | 12
Laceration (Injury, poisoning and procedural complications) | 4
Weight decreased (Investigations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 14
Back pain (Musculoskeletal and connective tissue disorders) | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Dizziness (Nervous system disorders) | 7
Headache (Nervous system disorders) | 11
Depression (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 17
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 23
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Blood blister (Skin and subcutaneous tissue disorders) | 6
Ecchymosis (Skin and subcutaneous tissue disorders) | 8
Petechiae (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 6
Haematoma (Vascular disorders) | 11
Hypertension (Vascular disorders) | 4

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed;

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial resul